CLINICAL TRIAL: NCT02405169
Title: Four Versus Six Endosseous Implants to be Used in the Rehabilitation of Totally Edentulous Patient in the Maxilla With Titanium Milled Framework
Brief Title: 4 vs 6 Implants in Totally Edentulous Patient in Maxilla With Ti. Cad-cam Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Franci (Other)
Responsible Party: Principal Investigator, Toia Marco, Four versus six endosseous implants to be used in the rehabilitation of totally edentulous patient in the maxilla with titanium milled framework: a randomized, controlled clinical trial., Institute Franci
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS-D-2012-031
Record Dates: First submitted 2015-03-16; First posted 2015-04-01 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Edentulous Maxilla
Keywords: Implantology; oral surgery; bone level changes; marginal bone level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test -4 implants- (Experimental): Evaluate marginal bone level (MBL) changes at implants that are placed in total edentulous patient when they are treated with four with titanium Cad/Cam framework.
  Interventions: Device: 4 vs 6 implant treatment in the maxilla
- Control -6 implants- (Active Comparator): Evaluate marginal bone level (MBL) changes at implants that are placed in total edentulous patient when they are treated with six with titanium Cad/Cam framework
  Interventions: Device: 4 vs 6 implant treatment in the maxilla

INTERVENTIONS:
Device: 4 vs 6 implant treatment in the maxilla
  Other Names: Astratech TX implant , Densply Implant (company name)

SUMMARY:
The primary objective of the present study is to evaluate the marginal bone level changes occurring in total edentulous patients treated with six or four implants.

Secondary objective

* overall survival rate
* soft tissue status by assessment of bleeding on probing (BoP) and probing pocket depth (PPD) at baseline and after 1,3,5 years
* prosthetic survival rates including screw or abutment loosening, framework or veneer fractures

DETAILED DESCRIPTION:
METHODS/PROCEDURES A randomized controlled multi-center clinical study is designed to determine whether a difference exists between the outcome of treatment when Astra tech implants are placed according to a six or a four implants protocol. The investigation will be performed in four centers: three in Italy affiliated to Institute Franci and one affiliated to the Department of Prosthodontics, Faculty of Odontology, Malmö University. In each center the clinician and the examiner will be the same person. The study protocol will be approved by the Regional Human Review Board of Padova General Hospital.

An investigators' meeting will be arranged prior to the starting with the patients' recruitment. Following a screening examination, subjects who will meet the inclusion criteria, will sign the Informed Consent and will be enrolled in the study. The period of patient enrollment will begin on January 1 2013 and ends December 31 2013.

The patients will be randomized with a method based on the use of sealed opaque envelopes. The cases will be assigned to two different treatment groups:

Group A- four implants (Test) Group B- six implants (Control)

Pre-treatment Patient data, medical history, clinical and radiographic examination will be recorded for each patient. Clinical photographs will be taken in frontal, occlusal and lateral projections.

Periodontal, endodontic and open caries lesions will be treated prior to implant installation. All patients will receive careful oral hygiene instructions and training in self-performed

plaque control measure. CT scan computed exams will be carried out. Plaster models and diagnostic wax-up will be carried out.

First Surgical Phase (Implant Installation) The patient will receive antibiotic prophylaxis (Amoxicillin 1gr) one hour prior to surgery and after the completion of implant installation until suture removal with 1gr three times a day. (If the patient is allergic to amoxicillin the examiner prescribes antibiotics at his own discretion at the same posology).

The surgical treatment will be performed under local anesthesia. In case of remaining teeth, they will be extracted with conventional technique before implants' placement. (13-14) Implants will be placed according to the guidelines described in the Astra Tech® manual "Surgical procedures", using a two-stage protocol.

Implant spinning during the positioning of the cover screw will be registered as positive, if present, or negative.

The operation will be finalized by a careful adaption of the flaps by means of an accurate suture in order to obtain a full periosteal coverage.

Intraoral clinical photographs before, during and after surgery will be taken.

Post-operative care The patients will be instructed to rinse with chlorhexidine 0.12% mouthrinse and will be told to rinse with the antiseptic solution three times a day for 2 weeks. The patients will be advised to take NSAIDs for pain relief at their own discretion.

Liquid and semisolid food will be prescribed for the first post-operative week, after which the sutures will be removed.

Two weeks after the operation the denture will be properly relined until the second stage surgery.

Patients will be controlled at third and sixth weeks.

Second surgical phase and Prosthetic procedures After eight weeks (+ 2) of healing in both groups (A and B) Uni Abutment 45° connection procedure will be performed. Impression with a customized spoon and Impregum material will be taken and the prosthetic procedure will be performed according to the Atlantis-Isus recommendations.

After 6 weeks (+ 2) from Uni Abutment connection the definitive full-arch fixed dental prostheses screw retained will be applied. The prosthesis will be made to accomplish the normal hygienic procedures. All prosthetic procedures will be made in accordance to the Astra Tech procedures & products manuals.

The length of bridge cantilevers will be duly calculated to minimize implant overloading according to the Atlantis-Isus recommendations (15)

Post-prosthetic measurements Clinical measurements Clinical examinations will be performed immediately following the installation of the definitive prosthesis (Baseline-Loading) and after 1, 3, and 5 years. In particular, plaque and soft-tissue inflammation will be registered. Clinical photographs will be taken at each interval point.

Plaque: the presence of plaque will be scored at each implant site as well as at level of the remaining teeth on four surfaces (buccal, lingual/palatal, mesial, distal). The mean percentage of plaque harboring surfaces will be calculated using the case as the unit.

Soft-tissue inflammation: the presence of soft-tissue inflammation (bleeding on probing) will be assessed on buccal, lingual/palatal, mesial, distal aspects of each implant. The mean percentage of inflamed sites will be calculated using the case as the unit.

Radiographic measurements Peri-apical radiographs will be taken at prosthesis insertion (Baseline) and after 1, 3, and 5 years.

The radiographs will be taken with an X-ray apparatus supplied with a long cone by the examiner each visiting time. Rinn centrators will be used to ensure reproducibility in the measurement of marginal bone level change.

The radiographic images will be analysed at the Department of Radiology of Sahlgrenska Academy, Gothenburg University by experienced radiologists who will be otherwise not involved in the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. age > 18 years;
2. edentulous maxilla or having hopeless remaining teeth that are intended to be extracted;
3. willingness to comply with all study requirements and to sign the IC;
4. have sufficient amount of bone (8mm or more) in the recipient site to allow implant placement without bone augmentation procedures.

Exclusion Criteria:

1. bone defects associated with severe knife-edge ridges;
2. bone defects resulting from tumor resection;
3. tobacco abuse (> 10 cigarettes/day);
4. severe kidney and liver disease;
5. history of radiotherapy in the head and neck region;
6. chemotherapy for treatment of malignant tumors at the time of the surgical procedure;
7. uncontrolled diabetes;
8. active periodontal disease involving the residual opposite dentition;
9. mucosal disease, such as lichen planus, in the areas to be treated;
10. poor oral hygiene;
11. non-compliant patients;
12. situations judged inconvenient(by the investigator) for the surgical treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Marginal bone resorption in millimeter from the the implant to the bone crest. | 1 year
Marginal bone resorption in millimeter from the the implant to the bone crest. | 3 year
Marginal bone resorption in millimeter from the the implant to the bone crest. | 5 year

SECONDARY OUTCOMES:
Fracture of the prosthetic components | 1 year
Fracture of the prosthetic components | 3 year
Fracture of the prosthetic components | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Denis Cecchinato, DDS, Study Director — Franci Institute
Locations (1):
- Franci Institute, Padua, Italy

REFERENCES:
- [Derived] Toia M, Moreira CS, Dias DR, Corra E, Ravida A, Cecchinato D. Fixed Full-Arch Maxillary Prostheses Supported by Four Versus Six Implants: 5-Year Results of a Multicenter Randomized Clinical Trial. Clin Oral Implants Res. 2025 Mar;36(3):298-313. doi: 10.1111/clr.14383. Epub 2024 Nov 24. PMID 39581887